CLINICAL TRIAL: NCT06422897
Title: Role of Anterior Segment Optical Coherence Tomography in Assessment of Healing of Thin or Perforated Cornea Treated by Amniotic Membrane Graft and Platelet Rich Plasma Clot
Brief Title: Role of AS-OCT in Assessment of Corneal Perforation
Acronym: OCT
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahemd Abdelghany, Associate professor, Minia University
Other Study IDs: 1133/04/2024
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Corneal Perforation
MeSH Terms: conditions — Corneal Perforation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cases after surgical management: cases are assessed by Anterior segment optical coherence tomography 1 month after surgical managemnt
  Interventions: Other: anterior segment optical coherence tomography

INTERVENTIONS:
Other: anterior segment optical coherence tomography — surgically treated corneal perforation by amniotic membrane graft and platelet rich plasma clot is assessed by anterior segment optical coherence tomography 1 month postoperative

SUMMARY:
Assessment of healing of thin and perforated cornea after surgical treatment by anterior segment optical coherence tomography

DETAILED DESCRIPTION:
* thin and perforated cornea (small perforation) is surgically treated by amniotic membrane graft and platelet rich plasma clot
* anterior segment optical coherence tomography is performed preoperative and 1 month postoperative to assess healing

ELIGIBILITY:
Inclusion Criteria:

* thin cornea about to perforate
* small corneal perforation

Exclusion Criteria:

* active infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients from both sexes was thin cornea or small corneal perforation surgically treated by amniotic membrane graft and platelet rich plasma clot
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Depth of corneal healing measured by optical coherence tomography | 1 month
  complete corneal healing by anterior segment optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Abdelghany, professor, Principal Investigator — professor
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abdelghany AA, Bahrawy ME, Alio JL. Combined Platelet Rich Plasma and Amniotic membrane in the treatment of Perforated Corneal Ulcers. Eur J Ophthalmol. 2022 Jul;32(4):2148-2152. doi: 10.1177/11206721211049100. Epub 2021 Oct 8. PMID 34623187